CLINICAL TRIAL: NCT01874743
Title: Pilot Study of the Impact of Rosuvastatin Administration on Residual Chronic Immune Activation Under Antiretroviral Therapy: CESAR (Crestor En Sus Des AntiRétroviraux)
Brief Title: Rosuvastatin to Decrease Residual Immune Activation in HIV Infection
Acronym: CESAR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut de Médecine et d'Epidémiologie Appliquée - Fondation Internationale Léon M'Ba (Other)
Collaborators: Sidaction (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: IMEA 043 CESAR
Record Dates: First submitted 2012-12-26; First posted 2013-06-11 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2012-12

CONDITIONS: HIV-1 Infection
Keywords: HIV,; Rosuvastatine,; Antiretroviral therapy
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rosuvastatine 20 mg (Experimental): Rosuvastatin 20 mg/day, once a day during 3 months
  Interventions: Drug: Rosuvastatin 20 mg/day

INTERVENTIONS:
Drug: Rosuvastatin 20 mg/day — All patients must take 20mg/day of rosavastatin during 3 months
  Other Names: Crestor ,(ZD 4522)

SUMMARY:
Participating countries: France Objectives Principal objective To evaluate, in HIV-1 infected patients receiving effective antiretroviral therapy, the effect of the addition of Rosuvastatin (dose of 20mg/day) for 3 months, on CD8 T cell activation as assessed by the proportion of peripheral CD8 T cells that co-express the activation markers CD38 and HLA-DR Secondary objectives To evaluate the effect of Rosuvastatin administration on residual CD4 and CD8 T cell activation To evaluate the effect of Rosuvastatin administration on the main serum soluble biomarkers of activation (CRP- HS, D-dimers, IL-6 and soluble CD14) To evaluate the effect of Rosuvastatin administration on CD4 T-cell count and on the CD4/CD8 T-cell ratio To study the relationship between the level of immune activation and the level of residual HIV replication in plasma To study the effect of Rosuvastatin administration on lipid profiles and the correlation between the HDL cholesterol and the CD4/CD8 T-cell ratio To evaluate the tolerance of Rosuvastatin at the dose of 20 mg/day

DETAILED DESCRIPTION:
Methodology Phase II pilot study; open-label; non comparative, bicentric, on-off design

Estimated enrolment 40 subjects

Outcomes Primary outcome :

• Variation at month 3 in the proportion of CD8 T lymphocytes co-expressing CD38 and HLA-DR

Secondary outcomes :

* Evolution of plasma/serum levels of CRP-HS, IL-6, soluble CD14 between baseline and month 3 and between month 3 and month 6
* Evolution of markers of CD4 T-cell activation (HLA-DR, Ki67) and CD8 T-cell activation (CD38, HLA-DR, Ki67) between baseline and month 3 and between month 3 and month 6 and evolution of the CD4/CD8 ratio between baseline and month 3 and between month 3 and month 6
* Evolution of CD4 T-cell count between baseline and month 3
* Evolution of HDL and LDL cholesterol between baseline and month 3 and between month 3 and month 6
* Relationship between HDL cholesterol and CD4/CD8 ratio at baseline, month 3 and month 6
* Relationship between the levels of T-cell activation and of plasma HIV-RNA levels at a detection level of 3 copies/mL
* Adverse events grade > 2 Eligibility Inclusion criteria
* HIV-infected patients receiving a combination of antiretroviral therapy for at least 24 months, unchanged since at least 18 months, exhibiting plasma HIV-RNA level below 20 copies and circulating CD4 T cell count below 500/mm3
* No indication for a treatment with statins (LDL cholesterol < 4.1 mmol/L under stable diet).

Non-inclusion criteria

* Patients receiving Maraviroc
* Patients receiving immune suppressing drugs
* Ongoing opportunistic, bacterial or viral infection
* CRP ≥ 10 mg/mL
* Co-infection with HCV (except if HCV cure), chronic HBV infection with active replication of HBV
* Indication for a treatment with statins
* Pregnancy
* CPK > 3x Normal values
* ALT or AST > 2x Normal values
* TG > 4 mmol/L
* DFG < 60 mL /min/1.73 m2
* Personal or familial history of genetic muscular disease
* History of muscular or hepatic toxicity with a statin or a fibrate
* Liver disease (TP < 70%).
* Hypothyroidism
* Concomitant treatment with : Kétoconazole, Itraconazole, Ciclosporine, Erythromycine, Cimétidine, Quinidine, Diltiazem, Vérapamil, systemic corticosteroids, Phénobarbital, Phénytoïne, Carbamazépine, Rifampicine, Lansoprazole
* Vaccination during the study

Intervention Rosuvastatin (20 mg/d per os) Intervention duration: 3 months Follow-up for 3 additional months

Statistical methods Bilateral Two-sided paired Wilcoxon to analyze the variation in the proportion of CD8 T lymphocytes that co-express CD38 and HLA-DR at month 3 (primary outcome).

The evolution of parameters of interest between 2 visits will also be analyzed using bilateral two-sided paired Wilcoxon test. Statistical significance will be considered for p< 0.05.

Substudies

Estimated planning or Study / Trial timetable Trial/study start date: April 2012 Enrolment period: 12 months Subject participation duration: 6 months Total trial/study duration: 18 months Estimated study/trial completion date: October 2013 [default date: date of last follow-up of last included patient, else justify the chosen date: date of "gel de la base de données", date of end of substudies analyses (think to delay for sampling transport, duration of technical analyses)]

Study / Trial design Phase II open-label pilot bicentric non comparative study. Patients eligible will receive Rosuvastatin for 3 months while continuing antiretroviral therapy. Patients will be followed-up 3 additional months after stopping the study drug (on-off design)

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected patients receiving a combination of antiretroviral therapy for at least 24 months, unchanged since at least 18 months, exhibiting plasma HIV-RNA level below 20 copies and circulating CD4 T cell count below 500/mm3
* No indication for a treatment with statins (LDL cholesterol < 4.1 mmol/L under stable diet).

Exclusion Criteria:

* Patients receiving Maraviroc
* Patients receiving immune suppressing drugs
* Ongoing opportunistic, bacterial or viral infection
* CRP ≥ 10 mg/mL
* Co-infection with HCV (except if HCV cure), chronic HBV infection with active replication of HBV
* Indication for a treatment with statins
* Pregnancy
* CPK > 3x Normal values
* ALT or AST > 2x Normal values
* TG > 4 mmol/L
* DFG < 60 mL /min/1.73 m2
* Personal or familial history of genetic muscular disease
* History of muscular or hepatic toxicity with a statin or a fibrate
* Liver disease (TP < 70%).
* Hypothyroidism
* Concomitant treatment with : Kétoconazole, Itraconazole, Ciclosporine, Erythromycine, Cimétidine, Quinidine, Diltiazem, Vérapamil, systemic corticosteroids, Phénobarbital, Phénytoïne, Carbamazépine, Rifampicine, Lansoprazole
* Vaccination during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
CD8 T cell activation | 6 months
  To evaluate, in HIV-1 infected patients receiving effective antiretroviral therapy, the effect of the addition of Rosuvastatin (dose of 20mg/day) for 3 months, on CD8 T cell activation as assessed by the proportion of peripheral CD8 T cells that co-express the activation markers CD38 and HLA-DR
Coexpress activation markers | 6 months
  proportion of peripheral CD8 T cells that co-express the activation markers CD38 and HLA-DR

SECONDARY OUTCOMES:
Rosuvastatin administration (on and off)on biomarkers activation | 6 months
  • Changes from baseline to month 3 (on rosuvastatin) and from month 3 to month 6 (off rosuvastatin) in levels of CRP-HS, IL-6, soluble CD14 Changes from baseline to month 3 (on rosuvastatin) and from month 3 to month 6 (off rosuvastatin) in the proportion of CD4 T cells expressing HLA-DR or Ki67 activation markers and in the proportion of CD8 T cells expressing HLA-DR and/or CD38 or Ki67 activation marker
Relationship between the levels of T-cell activation and of plasma HIV-RNA (ultrasensible measure) | 6 months
  • Relationship between the levels of T-cell activation and of plasma HIV-RNA levels at a detection level of 3 copies/mL
CD4 T-cell count and on the CD4/CD8 T-cell ratio | 6 months
  * Changes in CD4 T-cell count between baseline and month 3 •
  * Changes in the CD4/CD8 ratio between baseline and month 3 and between month 3 and month 6
Lipids profiles on and off rosuvastatine association | 6 months
  • Changes from baseline to month 3 (on rosuvastatin) and from month 3 to month 6 (off rosuvastatin) in levels of HDL and LDL cholesterol
Tolerance of Rosuvastatine | 6 months
  To evaluate the tolerance of Rosuvastatin at the dose of 20 mg/day (Number of patients with adverse events grade > 2)

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Weiss, PH,MD, Principal Investigator — HEGP
Locations (2):
- France (2):
  - St Antoine Hospital, Paris
  - HEGP, Paris